CLINICAL TRIAL: NCT01670448
Title: The Pectoral Nerve Block (PECBLOCK) for the Treatment of Pain After Breast Cancer Surgery.
Brief Title: PECBLOCK for the Treatment of Pain After Breast Surgery
Acronym: PECBLOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE12.231
Record Dates: First submitted 2012-08-17; First posted 2012-08-22 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2015-07

CONDITIONS: Cancer; Pain
Keywords: Postoperative pain; Chronic pain prevention; Regional anesthesia; Mastectomy
MeSH Terms: conditions — Neoplasms; Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PECBLOCK performed with bupivacaine (Active Comparator): Active drug given through PECBLOCK in these patients.
  Interventions: Procedure: PECBLOCK under echoguidance
- PECBLOCK performed with NaCl 0.9% (Placebo Comparator): Placebo drug given through PECBLOCK in these patients
  Interventions: Procedure: PECBLOCK under echoguidance

INTERVENTIONS:
Procedure: PECBLOCK under echoguidance — Performance of block under echography

SUMMARY:
Pain after breast cancer surgery could be severe and about 1/3 of patients will develop chronic pain. The PECBLOCK is the injection of local anesthetics between the two pectoral muscles to block pectoral nerves and intercostal nerves innervating the breast. The aim of this study is to evaluate the efficacy of the PECBLOCK performed under echoguidance in minor and major breast surgery. The prevention of chronic pain following surgery will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-85 yrs old
* patients ASA status I-IV

Exclusion Criteria:

* refusal of the PECBLOCK
* allergy to a drug used in the protocol (local anesthetic)
* patients with chronic pain before the surgery

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pain score at rest in the recovery room | 30 min after entering the recovery room or just before morphine administration if needed
  Using a 0-10 verbal numerical scale where 0 is no pain and 10 the worst pain imaginable

SECONDARY OUTCOMES:
Total morphine consumption in the recovery room | in the recovery room before discharge (after 1 h on average))
  When surgery is over and the patient is brought to the recovery room, the total morphine consumption in mg used in the recovery (for pain less than 4/10) is recorded

OTHER OUTCOMES:
Total sufentanil consumption during surgery | at the end of surgery (1-2 h on average)
  When surgery is over, 1-2 h on average depending if it is a tumorectomy or a mastectomy, the total sufentanil consumption in micrograms during surgery is recorded.
Assess any complication from PECBLOCK | first 24 hours post surgery
  Cardiovascular collapse, anaphylactic shock, hematoma, bleeding..?

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Cros, MD, Principal Investigator — CHU Limoges; Pierre Beaulieu, MD, Principal Investigator — CHUM
Locations (2):
- CHUM, Montreal, Quebec, Canada
- University Hospital, Limoges, Limoges, France

REFERENCES:
- [Derived] Cros J, Senges P, Kaprelian S, Desroches J, Gagnon C, Labrunie A, Marin B, Crepin S, Nathan N, Beaulieu P. Pectoral I Block Does Not Improve Postoperative Analgesia After Breast Cancer Surgery: A Randomized, Double-Blind, Dual-Centered Controlled Trial. Reg Anesth Pain Med. 2018 Aug;43(6):596-604. doi: 10.1097/AAP.0000000000000779. PMID 29672368